CLINICAL TRIAL: NCT03946423
Title: BAriaTric Surgery After Breast Cancer Treatment (BATS) - A Randomized Trial of Sleeve Gastrectomy Versus Lifestyle Intervention in Women Diagnosed With Early Stage Breast and With a BMI of ≥ 35
Brief Title: BAriaTric Surgery After Breast Cancer Treatment (BATS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018LS148
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Early-stage Breast Cancer; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve Gastrectomy & Lifestyle Intervention (Experimental)
  Interventions: Procedure: Bariatric Surgery with Sleeve Gastrectomy; Behavioral: Lifestyle Intervention
- Lifestyle Intervention (Active Comparator)
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Procedure: Bariatric Surgery with Sleeve Gastrectomy — Standard of care bariatric surgery with sleeve gastrectomy
  Arms: Sleeve Gastrectomy & Lifestyle Intervention
Behavioral: Lifestyle Intervention — All participants receive lifestyle intervention. The lifestyle intervention program is modeled closely after that used in the Diabetes Primary Prevention Trial and the LookAHEAD diabetes treatment studies. Intervention includes counseling sessions weekly for the first six months, twice a month during months 7-9, and monthly during months 10-12, and energy intake and exercise goal monitoring and guidance.

SUMMARY:
This is a feasibility study to gain an understanding of the willingness of women with a history of early stage breast cancer and current obesity to enroll in a weight-loss study, accept an assigned intervention (bariatric surgery with lifestyle intervention or lifestyle intervention alone), and comply with the study plan for 1 year. If there is successful enrollment in this study, the plan is to use what is learned in this study to design a larger, longer-term clinical trial to look at the effect of weight loss and incidence of cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer in the previous 10 years and currently disease free.
* Completion of breast cancer treatment (radiation, chemotherapy) at least > 6 months prior to enrollment
* Body mass index (BMI) of ≥ 35 kg/m2, but < 50 kg/m2.
* 18 through 67 years of age at enrollment
* Deemed healthy enough to undergo bariatric surgery, if assigned intervention, as determined by a surgeon and documented in the medical record.
* Must have insurance coverage with no exclusion for obesity related treatment or management of obesity related surgical complications - in general insurance coverage is available for persons with a BMI ≥ 35 kg/m2.
* Anticipated ability to abide by study requirements demonstrated in part by, but not limited to, successful completion of run-in assessments.
* Willingness to accept randomization into either interventional group.
* Provides voluntary written consent prior to performance of any research related activities.

Exclusion Criteria:

* Cardiovascular event (myocardial infarction, acute coronary syndrome, coronary artery angioplasty or bypass, stroke) in the past six months.
* Current evidence of congestive heart failure, angina pectoris, or symptomatic peripheral vascular disease.
* Cardiac stress test indicating that surgery or lifestyle would not be safe.
* 12-lead EKG indicating that surgery would not be safe.
* Significant anemia (hemoglobin 1.0 g/dL or more below normal range) or history of coagulopathy.
* History of stomach surgery, bile duct surgery, pancreatic surgery, splenectomy, or colon resection.
* Gastric or duodenal ulcer in the past six months.
* History of intra-abdominal sepsis except for uncomplicated appendicitis or diverticulitis more than six months prior to enrollment.
* Self-reported HIV-positive status, active tuberculosis, active malaria, chronic hepatitis B or C, cirrhosis, or inflammatory bowel disease.
* Currently pregnant or nursing, or planning to become pregnant in the next 15 months.
* History of alcohol, drug, or opioid dependency (excluding nicotine) in the past five years.
* Active psychosocial or psychiatric problem that is likely to interfere with adherence to the protocol.
* Deemed not an acceptable candidate by a trained psychologist.
* Current participation in a conflicting research protocol.
* Presence of any chronic or debilitating disease that would make adherence to the protocol difficult.
* Gastroesophageal reflux disease requiring medications. History of endoscopy demonstrating esophagitis or Barrett's changes in the esophagus.
* Any history of dysphagia.

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Weight Loss Intervention | 1 Year
  Feasibility for women who were diagnosed with early stage breast cancer in the previous 10 years and have a body mass index (BMI) of ≥ 35 kg/m2 but < 50 kg/m2.
Acceptability of Weight Loss Intervention | 1 Year
  Acceptability of women who were diagnosed with early stage breast cancer in the previous 10 years and have a body mass index (BMI) of ≥ 35 kg/m2 but < 50 kg/m2.

SECONDARY OUTCOMES:
Weight Loss | 1 Year
  Percent body mass weight loss
Breast Cancer Recurrence | 1 Year
  Incidence of breast cancer recurrence
Cancer Related Mortality | 1 Year
  Incidence of cancer related mortality
Overall Mortality | 1 Year
  Incidence of overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Anne Blaes, MD, Principal Investigator — University of Minnesota, Division of Hematology, Oncology and Transplantation